CLINICAL TRIAL: NCT00672685
Title: Assessment of the Efficacy of Omega-3 Fatty Acids Supplementation, Multi-domain Intervention or Their Combination on the Change of Cognitive Functions in Frail Elderly Subjects
Brief Title: Omega-3 Fatty Acids and/or Multi-domain Intervention in the Prevention of Age-related Cognitive Decline
Acronym: MAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 07 116 03
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Frail Elderly Subjects
Keywords: Cognitive decline; omega-3 fatty acids; nutrition; physical exercise; cognitive training; social activities; frailty
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity; Frailty | interventions — Docosahexaenoic Acids; Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Omega-3 group without any intervention
  Interventions: Dietary Supplement: omega-3
- 2 (Experimental): Omega-3 combined group (Omega-3 + multi-domain intervention)
  Interventions: Dietary Supplement: omega-3; Behavioral: multi-domain intervention
- 3 (Experimental): Placebo combined group (Placebo + multi-domain intervention)
  Interventions: Behavioral: multi-domain intervention; Drug: Placebo
- 4 (Placebo Comparator): Placebo group without any intervention
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: omega-3 — V0137 CA containing 400 mg docosahexaenoic acid (DHA) - 2 soft capsules once a day, i.e. 800 mg DHA per day for 36 months
  Other Names: Omega-3 fatty acids
  Arms: 1; 2
Behavioral: multi-domain intervention — multi-domain intervention = Nutrition, physical exercise, cognitive training and social activities, and preventive consultations
  Arms: 2; 3
Drug: Placebo — OMEGA-3 placebo
  Arms: 3; 4

SUMMARY:
Epidemiological and fundamental research carried out in recent years has highlighted the role played by omega-3 fatty acids in the process of cognitive decline that accompanies advancing age and Alzheimer's disease. In addition, it has been recognized for some years, following several convergent studies on the prevention of cognitive decline, that nutrition, physical exercise, cognitive training and social activities play a significant role in the maintenance of cognitive faculties. At present, there are a number of epidemiological arguments in favour of a protective role of each of these factors taken in isolation. It can be postulated that a multi-domain intervention may potentiate the protective role of omega-3 fatty acids.

The main objective of this study is to assess the efficacy of isolated supplementation with omega-3 fatty acid, an isolated multi-domain intervention (nutrition, physical exercise, cognitive stimulation, social activities), or their combination on the change of cognitive functions in frail elderly subjects aged of 70 years and older over 3 years.

Secondary objectives:

* To assess the efficacy of each treatment strategy on the change of functional capacities and the prevention of dependency,
* To study the long-term safety and tolerability of V0137,
* To study compliance and adhesion to the multi-domain intervention programme,

Ancillary studies :

To assess the impact of an intervention program on brain metabolism in FDG PET (MAPT-NI : : impact of multidomain intervention on brain metabolism (FDG-PET))

* To evaluate the impact of preventive strategies (Omega-3 treatment and multidomain intervention ) of MAPT study on brain atrophy (MRI),
* To evaluate the presence and density of ß-amyloid in MAPT subjects using AV45 PET scans (MAPT AV45),
* To determine if sleep disorders at early stage of Alzheimer 's disease could be predictive of cognitive decline and used as diagnosis tools (Mapt SLEEP)
* To evaluate the impact of omega-3 fatty acids on the body composition measured by DXA scans (MAPT-DXA)

DETAILED DESCRIPTION:
This is a multi-centre , randomised, placebo-controlled study in parallel groups in 1680 frail elderly subjects over the age of 70 years, living at home, monitored for a period of 3 years. The subjects will be randomised into one of the following 4 groups:

* Omega-3 group: 800 mg/day of docosahexaenoic acid (V0137CA nutritional supplement)
* Omega-3 + multi-domain intervention group: 800 mg/day of docosahexaenoic acid ( V0137CA)
* Placebo + multi-domain intervention group
* Placebo group The multi-domain intervention includes training / information sessions in the following 4 areas: nutrition, physical activity, cognitive training and social activities, and preventive consultations.

Selected subjects will present at least one of the following frailty criteria:

* Loss of one Instrumental Activity Daily Living (IADL)
* Subjective memory complaints to a physician
* Slow walking speed. Follow-up visits will occur every six months for 3 years for both dispensing of supplement and compliance (months 6, 12, 18, 24, 30 and 36) and neuropsychological and functional assessment (months 6, 12, 24, 36).

ELIGIBILITY:
Inclusion Criteria:

* subjects of both sex, aged of 70 years or over,
* subjects with at least one of the following frailty criteria: a subjective memory complaint, expressed to their attending physician, an inability to perform one of instrumental activities of daily living, a slow walking with a speed ≤ 0.77 m/s, i.e 5 seconds to walk 4 meters.
* subjects with an MMSE score of greater than or equal to 24,
* subjects capable of understanding the protocol, complying with its requirements and attending the study visits,
* subjects with sufficient availability to take part in the multi-domain intervention programme,
* subjects who, in the opinion of the investigator, are liable to comply with the treatment during the study;
* subjects capable of giving their written informed consent
* Covered by a health insurance system

Exclusion Criteria:

* Criteria related to diseases:

  * known presence of dementia or Alzheimer's disease (DSM IV criteria),
  * deterioration in global cognitive function (MMSE < 24),
  * dependency for basic activities of daily living (ADL<6),
  * presence of serious diseases, which could be life-threatening in the short term,
  * history or presence of any disease that could compromise the subject's participation in the multi-domain intervention sessions,
* Criteria related to treatments:

  o taking of supplements containing omega-3 (apart from food) within the past 6 months and/or taking omega-3 at inclusion.
* Criteria related to subjects:

  * visual or hearing impairments incompatible with performance and/or interpretation of the neuropsychological tests,
  * history or presence of any previous pathologies that could, in the opinion of the investigator, interfere with the results of the study or expose the subject to an additional risk,
  * subjects deprived of their freedom by administrative or judicial decision, or under guardianship or admitted to a healthcare or social institution,
  * participation in another clinical study in the previous month or participation scheduled during the study.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1680 (Actual)
Dates: Start 2008-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in cognitive function at 36 months determined by a composite score (sum of Z-score of 4 tests: FCRST test (free recall + total recall) score, MMSE orientation score, Wais-R score (Digit Substitution Symbol test), and the Category Naming Test score | Baseline, 6, 12, 24, 36 months

SECONDARY OUTCOMES:
Changes in other cognitive functions. Changes in functional capacities. To study the long-term safety and tolerability of V0137 CA treatment. To study compliance and adhesion to the "multi-domain" intervention program. | Baseline, 6, 12, 24, 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Vellas, MD-PhD, Principal Investigator — Toulouse University Hospital Centre
Locations (13):
- France (12):
  - University Hospital Bordeaux, Bordeaux
  - Regional Hospital, Castres
  - University Hospital of Dijon, Dijon
  - Regional Hospital, Foix
  - Regional Hospital, Lavaur
  - University Hospital Limoges, Limoges
  - UH of LYON SUD, Lyon
  - Chg Montauban, Montauban
  - University Hospital Montpellier, Montpellier
  - University Hospital of Nice, Nice
  - Regional Hospital, Tarbes
  - University Hospital Toulouse, Toulouse
- Princesse Grace Hospital, Monaco, Monaco

REFERENCES:
- [Derived] Coley N, Hoevenaar-Blom MP, Shourick J, van Charante EPM, van Dalen JW, van Gool WA, Richard E, Andrieu S; preDIVA study group and the MAPT/IHU HealthAge Open Science group. Searching for responders to multidomain dementia prevention in late life: A pooled analysis of individual participant data from the MAPT and preDIVA trials. Alzheimers Dement. 2025 Feb;21(2):e14472. doi: 10.1002/alz.14472. Epub 2025 Jan 17. PMID 39821948
- [Derived] de Assuncao Cortez Correa LC, Raffin J, Vellas B, Guerra RO, de Souto Barreto P. Sex-specific associations of neurodegeneration and inflammatory biomarkers with intrinsic capacity in older adults: Findings from the 4-year longitudinal Multidomain Alzheimer's Prevention Trial (MAPT). Maturitas. 2025 Feb;193:108191. doi: 10.1016/j.maturitas.2024.108191. Epub 2025 Jan 3. PMID 39754932
- [Derived] Aggarwal G, Morley JE, Vellas B, Nguyen AD, Butler AA; MAPT/DSA Group. Low circulating adropin concentrations predict increased risk of cognitive decline in community-dwelling older adults. Geroscience. 2024 Feb;46(1):897-911. doi: 10.1007/s11357-023-00824-3. Epub 2023 May 26. PMID 37233882
- [Derived] Giudici KV, de Souto Barreto P, Guyonnet S, Morley JE, Nguyen AD, Aggarwal G, Parini A, Li Y, Bateman RJ, Vellas B; MAPT/DSA Group. TNFR-1 and GDF-15 Are Associated With Plasma Neurofilament Light Chain and Progranulin Among Community-Dwelling Older Adults: A Secondary Analysis of the MAPT Study. J Gerontol A Biol Sci Med Sci. 2023 Mar 30;78(4):569-578. doi: 10.1093/gerona/glac244. PMID 36508390
- [Derived] Pages A, Costa N, Mounie M, Cestac P, De Souto Barreto P, Rolland Y, Vellas B, Molinier L, Juillard-Condat B; MAPT/DSA Group. Healthcare Costs Associated with Potentially Inappropriate Medication Prescribing Detected by Computer Algorithm Among Older Patients. Drugs Aging. 2022 May;39(5):367-375. doi: 10.1007/s40266-022-00938-x. Epub 2022 May 24. PMID 35606646
- [Derived] Rouch L, Rolland Y, Hanon O, Vidal JS, Cestac P, Sallerin B, Andrieu S, Vellas B, Barreto PS; MAPT/DSA Group. Blood pressure, antihypertensive drugs, and incident frailty: The Multidomain Alzheimer Preventive Trial (MAPT). Maturitas. 2022 Aug;162:8-14. doi: 10.1016/j.maturitas.2022.03.001. Epub 2022 Mar 15. PMID 35489133
- [Derived] Gonzalez-Bautista E, de Souto Barreto P, Salinas-Rodriguez A, Manrique-Espinoza B, Sourdet S, Rolland Y, Rodriguez-Manas L, Andrieu S, Vellas B; MAPT/DSA Group. Development and Validation of a Cutoff for the Chair Stand Test as a Screening for Mobility Impairment in the Context of the Integrated Care for Older People Program. J Gerontol A Biol Sci Med Sci. 2023 Jan 26;78(1):104-110. doi: 10.1093/gerona/glac055. PMID 35226732
- [Derived] Pages A, Costa N, Gonzalez-Bautista E, Mounie M, Juillard-Condat B, Molinier L, Cestac P, Rolland Y, Vellas B, De Souto Barreto P; MAPT/DSA Group. Screening for deficits on intrinsic capacity domains and associated healthcare costs. Arch Gerontol Geriatr. 2022 May-Jun;100:104654. doi: 10.1016/j.archger.2022.104654. Epub 2022 Feb 7. PMID 35193041
- [Derived] Raffin J, Angioni D, Giudici KV, Valet P, Aggarwal G, Nguyen AD, Morley JE, Guyonnet S, Rolland Y, Vellas B, de Souto Barreto P; MAPT/DSA Group. Physical Activity, Body Mass Index, and Blood Progranulin in Older Adults: Cross-Sectional Associations in the MAPT Study. J Gerontol A Biol Sci Med Sci. 2022 Jun 1;77(6):1141-1149. doi: 10.1093/gerona/glac018. PMID 35037052
- [Derived] He L, de Souto Barreto P, Sanchez Sanchez JL, Rolland Y, Guyonnet S, Parini A, Lucas A, Vellas B; MAPT/DSA Group. Prospective Associations of Plasma Growth Differentiation Factor 15 With Physical Performance and Cognitive Functions in Older Adults. J Gerontol A Biol Sci Med Sci. 2022 Dec 29;77(12):2420-2428. doi: 10.1093/gerona/glac020. PMID 35037034
- [Derived] Giudici KV, Guyonnet S, Morley JE, Nguyen AD, Aggarwal G, Parini A, Li Y, Bateman RJ, Vellas B, de Souto Barreto P; MAPT/DSA Group. Interactions Between Weight Loss and Plasma Neurodegenerative Markers for Determining Cognitive Decline Among Community-Dwelling Older Adults. J Gerontol A Biol Sci Med Sci. 2022 Jun 1;77(6):1159-1168. doi: 10.1093/gerona/glac015. PMID 35034116
- [Derived] Lu WH, Giudici KV, Rolland Y, Guyonnet S, Mangin JF, Vellas B, de Souto Barreto P. Associations Between Nutritional Deficits and Physical Performance in Community-Dwelling Older Adults. Front Nutr. 2021 Nov 11;8:771470. doi: 10.3389/fnut.2021.771470. eCollection 2021. PMID 34859035
- [Derived] Raffin J, Rolland Y, He L, Perus L, Mangin JF, Gabelle A, Virecoulon Giudici K, Vellas B, de Souto Barreto P; MAPT/DSA Group. Cross-sectional and longitudinal interaction effects of physical activity and APOE-epsilon4 on white matter integrity in older adults: The MAPT study. Maturitas. 2021 Oct;152:10-19. doi: 10.1016/j.maturitas.2021.06.010. Epub 2021 Jun 30. PMID 34674803
- [Derived] Costa N, Mounie M, Pages A, Derumeaux H, Rapp T, Guyonnet S, Coley N, Cantet C, Carrie I, Andrieu S, Molinier L. The Cost-Effectiveness of Three Prevention Strategies in Alzheimer's Disease: Results from the Multidomain Alzheimer Preventive Trial (MAPT). J Prev Alzheimers Dis. 2021;8(4):425-435. doi: 10.14283/jpad.2021.47. PMID 34585216
- [Derived] Coley N, Coniasse-Brioude D, Igier V, Fournier T, Poulain JP, Andrieu S; ACCEPT study group. Disparities in the participation and adherence of older adults in lifestyle-based multidomain dementia prevention and the motivational role of perceived disease risk and intervention benefits: an observational ancillary study to a randomised controlled trial. Alzheimers Res Ther. 2021 Sep 24;13(1):157. doi: 10.1186/s13195-021-00904-6. PMID 34560903
- [Derived] Conejero I, Dubois J, Gutierrez LA, Delrieu J, Arbus C, Garcia M, Lopez-Castroman J, Courtet P, Gabelle A. Amyloid Burden and Depressive Symptom Trajectories in Older Adults at Risk of Developing Cognitive Decline. J Clin Psychiatry. 2021 Aug 3;82(5):20m13410. doi: 10.4088/JCP.20m13410. PMID 34352166
- [Derived] Gonzalez-Bautista E, de Souto Barreto P, Andrieu S, Rolland Y, Vellas B; MAPT/DSA group (members are listed under 'Contributors'). Screening for intrinsic capacity impairments as markers of increased risk of frailty and disability in the context of integrated care for older people: Secondary analysis of MAPT. Maturitas. 2021 Aug;150:1-6. doi: 10.1016/j.maturitas.2021.05.011. Epub 2021 Jun 4. PMID 34274071
- [Derived] He L, de Souto Barreto P, Aggarwal G, Nguyen AD, Morley JE, Li Y, Bateman RJ, Vellas B; MAPT/DSA Group. Plasma Abeta and neurofilament light chain are associated with cognitive and physical function decline in non-dementia older adults. Alzheimers Res Ther. 2020 Oct 8;12(1):128. doi: 10.1186/s13195-020-00697-0. PMID 33032662
- [Derived] Gallini A, Yrondi A, Cantet C, Poncet M, Vellas B, Schmitt L, Andrieu S. Red Blood Cell Omega-3 Fatty Acid Composition and Psychotropic Drug Use in Older Adults: Results from the MAPT Study. J Nutr Health Aging. 2019;23(9):805-812. doi: 10.1007/s12603-019-1252-4. PMID 31641729
- [Derived] Guerville F, de Souto Barreto P, Taton B, Bourdel-Marchasson I, Rolland Y, Vellas B; Multidomain Alzheimer Preventive Trial (MAPT)/Data Sharing Alzheimer (DSA) Group. Estimated Glomerular Filtration Rate Decline and Incident Frailty in Older Adults. Clin J Am Soc Nephrol. 2019 Nov 7;14(11):1597-1604. doi: 10.2215/CJN.03750319. Epub 2019 Oct 18. PMID 31628118
- [Derived] Gabelle A, Gutierrez LA, Jaussent I, Navucet S, Grasselli C, Bennys K, Marelli C, David R, Andrieu S, Berr C, Vellas B, Dauvilliers Y. Excessive Sleepiness and Longer Nighttime in Bed Increase the Risk of Cognitive Decline in Frail Elderly Subjects: The MAPT-Sleep Study. Front Aging Neurosci. 2017 Sep 28;9:312. doi: 10.3389/fnagi.2017.00312. eCollection 2017. PMID 29033827
- [Derived] Andrieu S, Guyonnet S, Coley N, Cantet C, Bonnefoy M, Bordes S, Bories L, Cufi MN, Dantoine T, Dartigues JF, Desclaux F, Gabelle A, Gasnier Y, Pesce A, Sudres K, Touchon J, Robert P, Rouaud O, Legrand P, Payoux P, Caubere JP, Weiner M, Carrie I, Ousset PJ, Vellas B; MAPT Study Group. Effect of long-term omega 3 polyunsaturated fatty acid supplementation with or without multidomain intervention on cognitive function in elderly adults with memory complaints (MAPT): a randomised, placebo-controlled trial. Lancet Neurol. 2017 May;16(5):377-389. doi: 10.1016/S1474-4422(17)30040-6. Epub 2017 Mar 27. PMID 28359749
- [Derived] Gillette-Guyonnet S, Andrieu S, Dantoine T, Dartigues JF, Touchon J, Vellas B; MAPT Study Group. Commentary on "A roadmap for the prevention of dementia II. Leon Thal Symposium 2008." The Multidomain Alzheimer Preventive Trial (MAPT): a new approach to the prevention of Alzheimer's disease. Alzheimers Dement. 2009 Mar;5(2):114-21. doi: 10.1016/j.jalz.2009.01.008. PMID 19328438